CLINICAL TRIAL: NCT00634543
Title: Comparison of the Effectiveness and Safety Between Tramadol 37.5 Mg/Acetaminophen 325mg And Gabapentin for The Treatment of Painful Diabetic Neuropathy: Multicenter, Randomized, Open Comparative Study
Brief Title: A Study to Compare Safety and Efficacy of Tramadol Hydrochloride/Acetaminophen With Gabapentin in Participants With Diabetic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012967; ULT-KOR-06
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2013-07-16 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-07

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic neuropathy; Ultracet; Tramadol hydrochloride; Acetaminophen; Gabapentin
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Ultracet; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol hydrochloride (HCl)/ Acetaminophen (Experimental): Participants will receive 1 tablet containing tramadol HCl 37.5 milligram (mg) and acetaminophen 325 mg once daily, at bed time on Days 1 to 3, 1 tablet twice daily on Days 4 to 7 and 1 tablet thrice daily on Day 8 to 14. If there is no pain relief, the dosage can be increased up to 8 tablets per day for Days 15 to 28. The increased dose will be maintained for Days 29 to 42.
  Interventions: Drug: Tramadol hydrochloride/ Acetaminophen
- Gabapentin (Active Comparator): Participants will receive Gabapentin 300 mg once daily at bed time on Day 1, 300 mg twice daily on Day 2 and 300 mg thrice daily on Day 3. Gabapentin 300 mg will be administered twice daily (in the morning and midday) and gabapentin 600 mg in the evening on Day 8 to 14. If there is no pain relief, the dosage can be increased up to 3600 mg per day for Days 15 to 28. The increased dose will be maintained for Days 29 to 42.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Tramadol hydrochloride/ Acetaminophen — Participants will receive 1 tablet containing tramadol HCl 37.5 milligram (mg) and acetaminophen 325 mg once daily, at bed time on Days 1 to 3,. 1 tablet twice daily on Days 4 to 7 and 1 tablet thrice daily on Day 8 to 14. If there is no pain relief, the dosage can be increased up to 8 tablets per day for Days 15 to 28. The increased dose will be maintained for Days 29 to 42.
  Other Names: Ultracet
  Arms: Tramadol hydrochloride (HCl)/ Acetaminophen
Drug: Gabapentin — Participants will receive Gabapentin 300 mg once daily at bed time on Day 1, 300 mg twice daily on Day 2 and 300 mg thrice daily on Day 3. Gabapentin 300 mg will be administered twice daily (in the morning and midday) and gabapentin 600 mg in the evening on Day 8 to 14. If there is no pain relief, the dosage can be increased up to 3600 mg per day for Days 15 to 28. The increased dose will be maintained for Days 29 to 42.
  Arms: Gabapentin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of tramadol hydrochloride (HCl) 37.5 miligram (mg)/acetaminophen 325 mg compared to gabapentin in participants with diabetic neuropathic (nerve disorder caused by diabetes mellitus) pain.

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), multi-center and randomized (study drug is assigned by chance) study to compare the effectiveness and safety of tramadol HCl 37.5 mg/acetaminophen 325 mg with gabapentin in participants with diabetic neuropathy. The study will consist of 4 periods: Screening period (up to Day -14), Randomization period (Day 1), Dosage adjustment period (Day 15) and Maintenance period (Day 43). The participants will be randomly assigned to 1 of the 2 treatment groups: tramadol HCl 37.5 mg/acetaminophen 325 mg or gabapentin. Tramadol Hcl/acetaminophen group will receive 1 tablet for 3 days, then 1 tablet twice daily for 4 days followed by 1 tablet thrice daily for next 7 days. If there is no pain relief, the dosage can be increased up to 8 tablets per day for Day 15 to 28, and then the increased dosage will be maintained for Day 29 to 42. Gabapentin group will receive 300 mg on Day 1, 300 mg twice daily on Day 2, and 300 mg thrice daily for Day 3 to 7. Then for Day 8 to 14, participants will receive 300 mg in the morning, 300 mg in the midday and 600 mg in the evening. If there is no pain relief, gabapentin can be increased up to 3600 mg per day for Day 15 to 28, and then the increased dosage will be maintained for Day 29 to 42. Primarily, efficacy will be evaluated by pain intensity using numeric rating scale (NRS). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants having painful symmetric neuropathy (a disturbance in the function of the brain or spinal cord that may affect the nerves and muscles of the body) in the lower limbs applicable to both of the following conditions: decreased sensation of leg to monofilament, none or decreased ankle reflexes or decreased vibratory sensation and pain symptoms such as numbness (loss of sensation), tingling, paresthesia (a skin sensation, such as burning, prickling, itching, or tingling, with no apparent physical cause), burning, shooting pain, stabbing or lancinating (characterized by a sensation of cutting, piercing, or stabbing) pain
* Participants having painful diabetic neuropathy in the lower limbs for 3 months before randomization
* Participants diagnosed with Type ll diabetes and stable blood sugar level controlled with an oral medication, insulin or diet therapy for 3 months before randomization
* Participants with glycated hemoglobin (HbA1c) less than or equal to 10 percent
* Participants with pain intensity score of greater than or equal to 4 on numeric rating scale (NRS) for the last 48 hours

Exclusion Criteria:

* Participants who have previously experienced failure of tramadol treatment or have discontinued tramadol administration due to adverse event
* Participants who have received the prohibited medication before randomization (e.g., capsaicin, use of systemic steroids, steroid or local anesthetic injections, tramadol HCl or tramadol combination, gabapentin, opioid analgesics, antidepressants, anticonvulsants, alpha-lipoic acid, acupuncture, COX-2 selective inhibitors, long-acting NSAIDs, opioid analgesics, sedative-hypnotics, muscle relaxants, anxiolytics, antipsychotics, TENS, short-acting non-opioid analgesics)
* Participants with neuropathic pain caused by other reasons (e.g., alcohol abuse, connective tissue disease, toxic exposure, infection, neoplasm, ischemia)
* Participants suffering from painful diabetic neuropathy over 10 years
* Participants with physical damage or disease which may cause abnormal absorption, excessive accumulation, metabolism or excretion disorder of the study medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Hydrochloride/ Acetaminophen: Participants received 1 tablet containing tramadol hydrochloride (HCl) 37.5 milligram (mg) and acetaminophen 325 mg, once daily, at bed time on Day 1 to 3, 1 tablet twice daily on Day 4 to 7 and 1 tablet thrice daily on Day 8 to 14. If there was no pain relief, the dosage were increased up to 8 tablets per day for Day 15 to 28. The increased dose was maintained for Day 29 to 42.
- Gabapentin: Participants received gabapentin 300 mg once daily at bed time on Day 1, 300 mg twice daily on Day 2 and 300 mg thrice daily on Day 3. Gabapentin 300 mg was administered twice daily (in the morning and midday) and gabapentin 600 mg in the evening on Day 8 to 14. If there was no pain relief, the dosage were increased up to 3600 mg per day for Day 15 to 28. The increased dose was maintained for Day 29 to 42.
Period: Overall Study
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Started | 78 | 84
Treated | 76 | 80
Completed | 59 | 63
Not Completed | 19 | 21
Not completed — Other | 1 | 2
Not completed — Protocol Violation | 3 | 3
Not completed — Adverse Event | 11 | 11
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomly assigned participants who met the eligibility criteria and had at least 1 post-baseline efficacy assessment data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin | Total
Number analyzed (Participants) | 71 | 76 | 147
Age Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (7.4) | 56.6 (9.3) | 57.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 45 | 79
  Male | 37 | 31 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Intensity Score at Day 43
Description: Pain intensity was assessed on 11-point numerical rating scale ranging from 0=no pain to 10=pain as bad as you can imagine.
Time Frame: Baseline and Day 43
Population: Full analysis set (FAS) included all randomly assigned participants who met the eligiblility criteria and had at least 1 post-baseline efficacy assessment data. Last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Number analyzed (Participants) | 71 | 76
Units on a scale
  Baseline | 6.65 (1.60) | 6.30 (1.58)
  Change at Day 43 | 3.15 (1.83) | 2.76 (1.97)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride/ Acetaminophen vs Gabapentin; Test type: Non-Inferiority or Equivalence — Non inferiority was demonstrated if lower confidence limit of 2-sided 95% CI was less than the non-inferiority margin of 1.39; p = 0.2143, t-test, 2 sided; P-value was calculated for change from baseline in pain intensity score at Day 43; Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.23 to 1.01]

2. Secondary Outcome: Percentage of Participants With Pain Relief
Description: Pain relief was assessed on a scale ranging from -1 to 4, where -1=became worse, 0=no change, 1=relieved a little, 2=relieved moderately, 3=relieved a lot and 4=completely resolved.
Time Frame: Day 15, Day 29 and Day 43
Population: FAS included all randomly assigned participants who met the eligiblility criteria and had at least 1 post-baseline efficacy assessment data. Last observation carried forward (LOCF) was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Number analyzed (Participants) | 71 | 76
Percentage of Participants
  Day 15: Became worse | 1.4 | 4.0
  Day 15: No change | 12.7 | 14.5
  Day 15: Relieved a little | 31.0 | 34.2
  Day 15: Relieved moderately | 26.8 | 21.1
  Day 15: Relieved a lot | 26.8 | 26.3
  Day 15: Completely resolved | 1.4 | 0.0
  Day 29: Became worse | 4.2 | 1.3
  Day 29: No change | 9.9 | 10.5
  Day 29: Relieved a little | 25.4 | 29.0
  Day 29: Relieved moderately | 21.1 | 14.5
  Day 29: Relieved a lot | 38.0 | 44.7
  Day 29: Completely resolved | 1.4 | 0.0
  Day 43: Became worse | 2.8 | 1.3
  Day 43: No change | 7.0 | 11.8
  Day 43: Relieved a little | 22.5 | 25.0
  Day 43: Relieved moderately | 19.7 | 15.8
  Day 43: Relieved a lot | 46.5 | 42.1
  Day 43: Completely resolved | 1.4 | 4.0
Statistical Analysis 1: Comparison: Tramadol Hydrochloride/ Acetaminophen vs Gabapentin; Test type: Superiority or Other; p = 0.7539, Chi-squared; P-value was evaluated for pain relief in tramadol hydrochloride/ acetaminophen versus gabapentin groups at Day 15
Statistical Analysis 2: Comparison: Tramadol Hydrochloride/ Acetaminophen vs Gabapentin; Test type: Superiority or Other; p = 0.5905, Chi-squared; P-value was evaluated for pain relief in tramadol hydrochloride/ acetaminophen versus gabapentin groups at Day 29
Statistical Analysis 3: Comparison: Tramadol Hydrochloride/ Acetaminophen vs Gabapentin; Test type: Superiority or Other; p = 0.7407, Chi-squared; P-value was evaluated for pain relief in tramadol hydrochloride/ acetaminophen versus gabapentin groups at Day 43

3. Secondary Outcome: Overall Assessment of Study Medication by Participants
Description: Overall assessment of study medication was done by participants. Assessment was made on a scale of -2 to 2 where, -2=very bad, -1=bad, 0=no change, 1= good and 2=very good.
Time Frame: Day 43
Population: FAS included all randomly assigned participants who met the eligibility criteria and had at least 1 post-baseline efficacy assessment data. Here 'N' signifies number of participants who were evaluated for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Number analyzed (Participants) | 67 | 72
Percentage of participants
  Bad | 4.5 | 12.5
  No change | 29.9 | 29.2
  Good | 50.8 | 41.7
  Very good | 14.9 | 16.7
Statistical Analysis 1: Comparison: Tramadol Hydrochloride/ Acetaminophen vs Gabapentin; Test type: Superiority or Other; p = 0.3504, Chi-squared; P-value was evaluated for all categories (bad, no change, good and very good)

4. Secondary Outcome: Overall Assessment of Study Medication by Investigator
Description: Overall assessment of study medication was done by Investigator. Assessment was made on a scale of -2 to 2 where, -2=very bad, -1=bad, 0=no change, 1= good and 2=very good.
Time Frame: Day 43
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Number analyzed (Participants) | 67 | 72
Percentage of participants
  Bad | 0 | 2.8
  No change | 31.3 | 30.6
  Good | 50.8 | 51.4
  Very good | 17.9 | 15.3
Statistical Analysis 1: Comparison: Tramadol Hydrochloride/ Acetaminophen vs Gabapentin; Test type: Superiority or Other; p = 0.5690, Chi-squared; P-value was evaluated for all categories (bad, no change, good and very good)

5. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Score at Day 43
Description: The BPI is a questionnaire designed to assess the severity and impact of pain on quality of life. Pain severity score is caculated by sum of all severity items (pain worst, pain least, pain average and pain now) divided by pain now. Total score for pain severity ranges from 0=no pain to 10=extreme pain. Pain interference score was calculated by sum of all interference items (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life) score. Total score for pain interference ranges from 0=no interference to 70= interferes completely.
Time Frame: Baseline and Day 43
Population: FAS included all randomly assigned participants who met the eligibility criteria and had at least 1 post-baseline efficacy assessment data. Here 'n' signifies number of participants who were evaluated for this outcome measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Number analyzed (Participants) | 71 | 76
Units on a scale
  Baseline: Pain severity score (n=68, 73) | 4.5 (1.3) | 4.9 (1.8)
  Change at Day 43: Pain severity score (n=60, 60) | 0.1 (2.3) | 0.1 (1.9)
  Baseline: Pain interference score (n=71, 76) | 30.2 (14.8) | 29.8 (14.8)
  Change at Day 43:Pain interference score(n=63, 68) | -11.0 (15.4) | -8.8 (14.7)

6. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Score at Day 43
Description: The SF-36 is designed to assess the health status of participants. The SF-36 includes 1 multi-item scale measuring physical health and mental health. Physical health includes physical functioning, role limitations due to physical health, pain and general health. Mantal health includes role limitations due to emotional problems, energy/fatigue, emotional well being and social functioning. Each item is scored on a 0-100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state.
Time Frame: Baseline and Day 43
Population: FAS included all randomly assigned participants who met the eligibility criteria and had at least 1 post-baseline efficacy assessment data. Here 'n' signifies number of participants who were evaluated for at given time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Number analyzed (Participants) | 71 | 76
Units on a scale
  Baseline: Phiysical functioning (n=71,76) | 56.3 (24.1) | 60.6 (24.5)
  Change at Day 43: Physical functioning (n=63, 68)) | 3.2 (19.7) | 3.2 (19.4)
  Baseline: Physical role limitation (n=71,76) | 42.3 (42.8) | 49.3 (41.6)
  Change at Day 43:Physical role limitation(n=62,68) | 13.7 (41.4) | 10.7 (43.3)
  Baseline: Pain (n=71,76) | 49.3 (20.9) | 50.8 (18.1)
  Change at Day 43: Pain (n=63, 68) | 15.6 (22.7) | 10.4 (22.2)
  Baseline: General health (n=71,76) | 38.0 (20.4) | 40.3 (17.8)
  Change at Day 43: General health (n=63, 68) | 4.6 (18.8) | 4.4 (14.1)
  Baseline: Emotional role limitation (n=71,76) | 46.9 (44.9) | 50.4 (45.7)
  Change at Day43:Emotional role limitation(n=63,68) | 12.7 (49.9) | 18.1 (47.3)
  Baseline: Energy/Fatigue (n=71,76) | 39.4 (22.1) | 42.6 (19.7)
  Change at Day 43: Energy/Fatigue (n=63, 68) | 5.7 (21.8) | 10.0 (17.8)
  Baseline: Emotional well-being (n=71,76) | 57.2 (22.0) | 61.4 (18.9)
  Change at Day 43: Emotional well being (n=63, 68) | 5.3 (23.3) | 7.0 (16.0)
  Baseline: Social functioning (n=71,76) | 68.3 (23.3) | 72.2 (24.5)
  Change at Dya 43: Social functioning (n=63, 68) | 9.9 (24.9) | 5.5 (24.9)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 43
Description: Safety analysis population included all randomly assigned participants who received at least 1 dose of study medication.
Arm/Group | Tramadol Hydrochloride/ Acetaminophen | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/80
Other Adverse Events (participants affected / at risk) | 33/76 | 18/80
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride/ Acetaminophen (N=76) | Gabapentin (N=80)
Dizziness (Nervous system disorders) | 13 | 10
Somnolence (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 14 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 3

LIMITATIONS AND CAVEATS:
The study was a non-inferiority study to demonstrate that tramadol/acetaminophen did not have poorer ffectiveness as compared to gabapentin. However this could not be demonstrated because of error in the minimum significant difference set-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is cancelled.